CLINICAL TRIAL: NCT00316095
Title: Reduced Factorial Design, Randomized, Double Blind Trial Comparing Combinations of Telmisartan 20 or 80 mg and Simvastatin 20 or 40 mg With Single Component Therapies in the Treatment of Hypertension and Dyslipidemia
Brief Title: Combination of Telmisartan and Simvastatin in the Treatment of Hypertension and Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1228.1; EudraCT No.: 2005-002851-41
Record Dates: First submitted 2006-04-19; First posted 2006-04-20 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Telmisartan; Simvastatin

INTERVENTIONS:
Drug: telmisartan
Drug: simvastatin

SUMMARY:
This study will investigate two registered drugs, one for the treatment of high blood pressure and one for the treatment of elevated cholesterol. High blood pressure (hypertension) is a common medical condition affecting millions of people worldwide. A wide variety of effective drug treatments is available to reduce blood pressure. Elevated cholesterol (hypercholesterolemia) is a common medical condition affecting people worldwide. A wide variety of effective drug treatments is available to reduce cholesterol levels.

Hypertension and hypercholesterolemia often occur together. They are both important risk factors for the development of heart and vessel diseases (e.g. heart attack or stroke). Current guidelines advise treatment of high blood pressure and elevated cholesterol to reduce the risk of cardiovascular diseases. This study will test the simultaneous use of a drug to reduce blood pressure and a drug to reduce elevated cholesterol. Both drugs are registered and are effective. The drug for treatment of high blood pressure is telmisartan Micardis). The drug for treatment of elevated cholesterol is simvastatin (Zocor). Since hypertension and hypercholesterolemia frequently occur together, the purpose of this study is to investigate whether both drugs can be used simultaneously. A low dose and a high dose of these drugs will be used. It will be investigated whether each of the drugs is still as effective when given together, at the same time of day, with the other drug.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Age 18 years or older
* Hypertension as defined by a mean seated cuff DBP of >=95 - 109 mmHg
* Hypercholesterolemia as defined by a fasting LDL-C level at visit 2 according to
* CV risk shown in table below:

  * CV Risk Group:

    1. Group I Hypertension and Hypercholesterolemia only
    2. Group II Hypertension and Hypercholesterolemia plus > 1 risk factors
    3. Group III Hypertension and Hypercholesterolemia plus CHD and/or diabetes mellitus and/or other athero-sclerotic disease
* Fasting LDL-C group I and II: 100-250 mg/dL (2.6-6.5 mmol/L)
* Fasting LDL-C group III: 100-160 mg/dL (2.6-4.1 mmol/L)
* Risk factors: >= 45 yrs if male, >= 55 years if female, family history of CHD, current smoker, HDL-C < 40 mg/dL

Exclusion Criteria:

* pre-menopausal women who are not surgically sterile or are nursing or pregnant or are of child-bearing potential and are not practicing acceptable means of birth control
* inability to stop current antihypertensive and/or cholesterol-lowering therapies
* contraindication to a washout/placebo treatment
* clinically relevant cardiac arrhythmias
* hypertrophic obstructive cardiomyopathy, hemodynamically relevant stenosis of the aortic or mitral valve
* mean sitting SBP >=180 mmHg or mean sitting DBP >=110 mmHg at two consecutive visits
* known or suspected secondary hypertension
* known or suspected secondary hyperlipidemia of any etiology
* diabetes that has not been stable and controlled for the previous three months
* severe renal dysfunction
* bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post-renal transplant or one kidney
* biliary obstructive disorders, hepatic insufficiency, including past or current liver disease
* clinically relevant hypokalaemia or hyperkalaemia
* uncorrected volume depletion
* uncorrected sodium depletion
* any history of myopathy or rhabdomyolysis during the past treatment with HMG Co-A reductase inhibitors
* concurrent use of large quantities of grapefruit juice
* known hypersensitivity or intolerance to HMG Co-A reductase inhibitors and/or angiotensin receptor blockers, hereditary fructose intolerance
* planned significant diet and/or lifestyle (including exercise) changes during the treatment phase of the trial
* history of drug or alcohol dependency
* any investigational drug therapy within one month of providing informed consent
* any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of the trial medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1695
Dates: Start 2006-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08

PRIMARY OUTCOMES:
Change in 24-hour ambulatory blood pressure measurement (ABPM) measured mean diastolic blood pressure (DBP) | 8 weeks
Change in 24-hour ambulatory blood pressure measurement (ABPM) measured mean low density lipoprotein (LDL) | 8 weeks

SECONDARY OUTCOMES:
Change in the 24-hour ABPM (Ambulatory Blood Pressure Monitoring) measured mean SBP | after 8 weeks
Changes in Trough-to-peak ratios of SBP and DBP, taken from ABPM | after 8 weeks
Changes in Seated morning DBP and SBP | after 8 weeks
Response rate to blood pressure treatment | after 8 weeks
Response rate to lipid lowering treatment | after 8 weeks
Change in Total cholesterol | after 8 weeks
Change in HDL-cholesterol | after 8 weeks
Change in triglycerides | after 8 weeks
Change in Apolipoprotein B | after 8 weeks
Change in free fatty acids | after 8 weeks
Change in Adiponectin | after 8 weeks
Change in HOMA-index | after 8 weeks
Change in haemoglobin A1C | after 8 weeks
Changes in high sensitive c-reactive protein | after 8 weeks
Changes in microalbuminuria | after 8 weeks
Adverse events | up to 15 weeks
Changes in clinical laboratory parameter | up to 15 weeks
Assessment of pulse rate | up to 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim BV/Alkmaar
Locations (77):
- Czechia (8):
  - Boehringer Ingelheim Investigational Site, Benátky nad Jizerou
  - Boehringer Ingelheim Investigational Site, Brno
  - Boehringer Ingelheim Investigational Site, Mladá Boleslav
  - Boehringer Ingelheim Investigational Site, Pilsen
  - Boehringer Ingelheim Investigational Site, Prague
  - Boehringer Ingelheim Investigational Site, Příbram
  - Boehringer Ingelheim Investigational Site, Uničov
  - Boehringer Ingelheim Investigational Site, Ústí nad Orlicí
- France (4):
  - ALTI, Angers
  - Boehringer Ingelheim Investigational Site, Angers
  - Boehringer Ingelheim Investigational Site, Sidi Daoud Tunis
  - Boehringer Ingelheim Investigational Site, Tunis
- Germany (9):
  - Boehringer Ingelheim Investigational Site, Haag
  - Boehringer Ingelheim Investigational Site, Mainz
  - Boehringer Ingelheim Investigational Site, Neuburg A. D. Donau
  - Boehringer Ingelheim Investigational Site, Nuremberg
  - Boehringer Ingelheim Investigational Site, Rednitzhembach
  - Boehringer Ingelheim Investigational Site, Unterschneidheim
  - Boehringer Ingelheim Investigational Site, Westerkappeln
  - Boehringer Ingelheim Investigational Site, Wiesbaden
  - Boehringer Ingelheim Investigational Site, Würzburg
- Boehringer Ingelheim Investigational Site, Hong Kong, Hong Kong
- Netherlands (15):
  - Boehringer Ingelheim Investigational Site, Almere Stad
  - Boehringer Ingelheim Investigational Site, Beek en Donk
  - Andromed Breda, Breda
  - Gemini Ziekenhuis, Den Helder
  - Andromed Eindhoven, Eindhoven
  - Boehringer Ingelheim Investigational Site, Ewijk
  - Andromed Noord, Groningen
  - Andromed Leiden, Leiden
  - Andromed Nijmegen, Nijmegen
  - Boehringer Ingelheim Investigational Site, Oude Pekela
  - Andromed Rotterdam, Rotterdam
  - Julius Center for Patient oriented Research, Utrecht
  - Andromed Oost, Velp
  - Boehringer Ingelheim Investigational Site, Wildervank
  - Andromed Zoetermeer, Zoetermeer
- Russia (2):
  - Boehringer Ingelheim Investigational Site, Moscow
  - Boehringer Ingelheim Investigational Site, Saint Petersburg
- Slovakia (9):
  - Boehringer Ingelheim Investigational Site, Bratislava
  - Boehringer Ingelheim Investigational Site, Košice
  - Boehringer Ingelheim Investigational Site, Kralovsky Chmlec
  - Boehringer Ingelheim Investigational Site, Liptovský Hrádok
  - Boehringer Ingelheim Investigational Site, Nitra
  - Boehringer Ingelheim Investigational Site, Považská Bystrica
  - Boehringer Ingelheim Investigational Site, Prešov
  - Boehringer Ingelheim Investigational Site, Trenčín
  - Boehringer Ingelheim Investigational Site, Vráble
- South Africa (6):
  - Boehringer Ingelheim Investigational Site, Boksburg
  - Boehringer Ingelheim Investigational Site, Cape Town
  - Boehringer Ingelheim Investigational Site, Durban
  - Boehringer Ingelheim Investigational Site, Johannesburg
  - Boehringer Ingelheim Investigational Site, Krugersdorp
  - Boehringer Ingelheim Investigational Site, Midrand
- South Korea (6):
  - Chonnam National University Hospital, Kwangju
  - Hallym University Sacred Heart Hospital, Kyunggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Korea University Medical Center, Seoul
  - St. Mary Hospital, Seoul
- Sweden (7):
  - Medicinkliniken, Gothenburg
  - Medicinkliniken, Lule?
  - Boehringer Ingelheim Investigational Site, Lule?
  - Endokrinologkliniken, Malmo
  - Boehringer Ingelheim Investigational Site, Rättvik
  - Medicinkliniken, Stockholm
  - Boehringer Ingelheim Investigational Site, Uppsala
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Ukraine (7):
  - Boehringer Ingelheim Investigational Site, Dnipro
  - Boehringer Ingelheim Investigational Site, Ivano-Frankivsk
  - Boehringer Ingelheim Investigational Site, Kharkiv
  - Boehringer Ingelheim Investigational Site, Kiev
  - Boehringer Ingelheim Investigational Site, Lutsk
  - Boehringer Ingelheim Investigational Site, Lviv
  - Boehringer Ingelheim Investigational Site, Zaporizhzhya